CLINICAL TRIAL: NCT00860717
Title: Clinic-Epidemiological Evaluation of Ulcers in Leprosy Patients and the Use of Low Level Laser Therapy: a Randomized Clinical Trial
Brief Title: The Use of Low Level Laser Therapy for Wound Healing in Leprosy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Para Federal University (Other)
Responsible Party: Claudio Guedes Salgado, Federal University of Pará
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FINEP 1460/03
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-03

CONDITIONS: Leprosy
Keywords: Leprosy; Ulcers; Laser
MeSH Terms: conditions — Leprosy; Ulcer | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects from the arm number 1 received routine treatment, including daily simple dressings with sterile gauze after wound cleaning with a 0.9% physiologic solution, use of 1% hydrophilic silver sulfadiazine cream (Prati Donaduzzi Laboratory, Toledo, Brazil) and orientation about the use of adapted footwear, self-care and the prevention of disabilities. Surgical debridement was done whenever indicated by nursing or orthopedic services from UREMC.
  Interventions: Procedure: Routine treatment
- 2 (Experimental): Subjects from the arm number 2 received low level laser therapy 3 times per week for 12 weeks, in addition to the same treatment as patients from the arm number 1.
  Interventions: Radiation: Low level laser therapy (LLLT)

INTERVENTIONS:
Procedure: Routine treatment — Subjects from the Control Group received routine treatment, including daily simple dressings with sterile gauze after wound cleaning with a 0.9% physiologic solution, use of 1% hydrophilic silver sulfadiazine cream (Prati Donaduzzi Laboratory, Toledo, Brazil) and orientation about the use of adapted footwear, self-care and the prevention of disabilities. Surgical debridement was done whenever indicated by nursing or orthopedic services from UREMC.
  Arms: 1
Radiation: Low level laser therapy (LLLT) — The LLLT equipment was an indium-gallium-aluminnium-phosphide (InGaAlP) semiconductor laser with a maximum output power of 40 mW, continuous radiation emission of visible red light with 660 nm wavelength (+/- 10 nm) and a spot area of 0.04 cm². The energy density used was 4 J per point in the wound edges and 2 J/cm² in the wound bed with a power density of 1 W/cm2.
  Wound beds were irradiated using a scanning technique with no direct contact.
  Other Names: LLLT; Cold laser; LILT
  Arms: 2

SUMMARY:
Neuropathic ulcers are common sequelae of leprosy. The objectives of this study are to analyze the clinic-epidemiological characteristics of patients attended at one specialized dressing service from a leprosy-endemic region of the Brazilian Amazon and to evaluate the effect of Low Level Laser Therapy on wound healing of these patients.

ELIGIBILITY:
Inclusion Criteria:

* presented with neuropathic ulcer
* attended at least 3 weekly appointments at the dressing service of UREMC
* completed specific multi-drug therapy for M. leprae
* gave written informed consent to participate in the study

Exclusion Criteria:

* clinically detectable infection in the ulcer
* use of drugs, like corticosteroids that could interfere with the wound healing process
* use of special dressings like hydrocolloid, calcium alginate, activated carbon or any kind of therapeutic procedure different from that used routinely for both groups of study
* non-attendance to therapeutic program (six sequential times or nine intercalated)
* pregnancy
* discomfort during treatment procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Wound healing | Biweekly until the end of the 12 week treatment period.

SECONDARY OUTCOMES:
Ulcer surface area, depth and PUSH tool score. | Biweekly until the end of the 12 week treatment period or until complete cicatrization of the treated ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G Salgado, Dr, Study Director — Federal University of Pará
Locations (1):
- Dr. Marcello Candia Reference Unit in Sanitary Dermatology of the State of Pará in Brazil (UREMC), Marituba, Pará, Brazil

REFERENCES:
- [Background] Flemming K, Cullum N. Laser therapy for venous leg ulcers. Cochrane Database Syst Rev. 2000;(2):CD001182. doi: 10.1002/14651858.CD001182. PMID 10796615
- [Background] Hopkins JT, McLoda TA, Seegmiller JG, David Baxter G. Low-Level Laser Therapy Facilitates Superficial Wound Healing in Humans: A Triple-Blind, Sham-Controlled Study. J Athl Train. 2004 Sep;39(3):223-229. PMID 15496990
- [Background] Schindl A, Schindl M, Pernerstorfer-Schon H, Mossbacher U, Schindl L. Low intensity laser irradiation in the treatment of recalcitrant radiation ulcers in patients with breast cancer--long-term results of 3 cases. Photodermatol Photoimmunol Photomed. 2000 Feb;16(1):34-7. doi: 10.1034/j.1600-0781.2000.160109.x. PMID 10721863
- [Background] Lucas C, van Gemert MJ, de Haan RJ. Efficacy of low-level laser therapy in the management of stage III decubitus ulcers: a prospective, observer-blinded multicentre randomised clinical trial. Lasers Med Sci. 2003;18(2):72-7. doi: 10.1007/s10103-003-0259-5. PMID 12928815
- [Background] Franek A, Krol P, Kucharzewski M. Does low output laser stimulation enhance the healing of crural ulceration? Some critical remarks. Med Eng Phys. 2002 Nov;24(9):607-15. doi: 10.1016/s1350-4533(02)00112-1. PMID 12376047
- [Background] Schubert V. Effects of phototherapy on pressure ulcer healing in elderly patients after a falling trauma. A prospective, randomized, controlled study. Photodermatol Photoimmunol Photomed. 2001 Feb;17(1):32-8. doi: 10.1034/j.1600-0781.2001.017001032.x. PMID 11169174
- [Background] Pereira AN, Eduardo Cde P, Matson E, Marques MM. Effect of low-power laser irradiation on cell growth and procollagen synthesis of cultured fibroblasts. Lasers Surg Med. 2002;31(4):263-7. doi: 10.1002/lsm.10107. PMID 12355572
- [Derived] Barreto JG, Salgado CG. Clinic-epidemiological evaluation of ulcers in patients with leprosy sequelae and the effect of low level laser therapy on wound healing: a randomized clinical trial. BMC Infect Dis. 2010 Aug 10;10:237. doi: 10.1186/1471-2334-10-237. PMID 20698989